CLINICAL TRIAL: NCT02116712
Title: The Tolerability of Saracatinib in Subjects With Lymphangioleiomyomatosis (LAM) (SLAM-1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tony Eissa (Other)
Collaborators: University of Texas (Other); University of Cincinnati (Other)
Responsible Party: Sponsor-Investigator, Tony Eissa, Professor of Medicine - Pulmonary, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLAM 7601
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Pulmonary Lymphangioleiomyomatosis
Keywords: LAM; saracatinib; Lymphangioleiomyomatosis
MeSH Terms: conditions — Lymphangioleiomyomatosis | interventions — saracatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Saracatinib (Experimental): Only one arm: Intervention is Saracatinib. We plan to study three escalating doses of oral saracatinib; 50, 125 and 175 mg. Saracatinib is given orally once a day.
  More regarding dose escalation is included in intervention below.
  Interventions: Drug: Saracatinib

INTERVENTIONS:
Drug: Saracatinib — Saracatinib is escalated as follows: Three dose levels will be administered for 1 month each: 50 mg, 125 mg and 175 mg. Three subjects will be treated at the lowest daily dose of 50 mg. If no subject experiences DLT (dose limiting toxicity), the dose level is escalated to 125 mg/day for the next cohort of 3 different subjects and so on to next dose.
  Other Names: AZD0530

SUMMARY:
Lymphangioleiomyomatosis (LAM) is a rare lung disease that mostly affects women of childbearing age. In LAM, abnormal, muscle-like cells begin to grow out of control in the lungs. As a result, air can't move freely in and out of the lungs. In some cases, this means the lungs can't supply the body's other organs with enough oxygen.

This study is being conducted to find out what dose of a drug called saracatinib is best tolerated by people with LAM. This drug has been tested in patients with certain types of cancer but is not currently approved by the United States Food and Drug Administration (FDA). Saracatinib may work in cancer by preventing the growth, movement and invasiveness of cancer cells. The use of saracatinib to treat LAM is considered experimental. Preliminary testing already completed suggests that the study drug, saracatinib, may suppress certain substances in the lungs of patients with LAM thus may be effective in slowing down the disease process

DETAILED DESCRIPTION:
Tuberous sclerosis complex (TSC) is an autosomal dominant disorder caused by mutations in tuberous sclerosis complex 1 (TSC1) or tuberous sclerosis complex 2 (TSC2) tumor suppressor genes. TSC is characterized by tumors in a wide range of tissues, seizures, mental retardation, autism, and organ failure. Lymphangioleiomyomatosis (LAM), the major pulmonary manifestation in women with TSC, is a progressive lung disease characterized by infiltration of atypical smooth muscle like cells and formation of cysts.

The long term goal of this research is to devise novel therapeutic strategies for patients with LAM. Our preliminary data reveal an increase in active Src in lung tissues of patients with LAM as well as in laboratory cultured cells.

The focus of this study is to examine if Src inhibition represents a potential therapeutic strategy in LAM. In this study, we will evaluate the safety, tolerability of Src inhibition in subjects with LAM.

The Quality Assurance (QA) plan is put forth in the Manual of Operations for this study. This study is utilizing the services of the Data Coordinating Center (DCC) at the University of Southern Florida. The data collected and entered in the electronic clinical research form (CRF) at each site will be reviewed by the site clinical research associate and the DCC data manager. Data check will be made throughout the study for all 3 sites and for all patients enrolled. Data checks to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry.

Source data verification will be done to assess the accuracy, completeness, or representativeness of registry data. This will be done by a DCC Clinical Research Associate (CRA).

Each site has received a copy of the general Manual of Operations, the Pharmacy Manual of Operations and the Laboratory Manual of Operations. Standard Operating Procedures to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management.

We will apply the standards set forth in the National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE)version V 4.0.

Adverse events related to study medication will be tabulated by body system and by severity using the NCI CTCAE v4.0. A dose-limiting toxicity (DLT) is defined as any CTCAE grade ≥3 toxicity despite adequate treatment and considered by the investigator to be possibly related to saracatinib treatment. A grade 3 adverse event is defined as severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care.

Adverse events related to study medication will be tabulated by body system and by severity using the NCI CTCAE v4.0. A dose-limiting toxicity (DLT) is defined as any CTCAE grade ≥3 toxicity despite adequate treatment and considered by the investigator to be possibly related to saracatinib treatment. A grade 3 adverse event is defined as severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care. Below are some examples of what would be considered DLT. Other grade 3 events will be evaluated by investigator on a case-by-case basis to determine if they are drug related.

1. Allergic reaction: Prolonged (e.g., not rapidly responsive to symptomatic medication; recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates)
2. Anaphylaxis: Symptomatic bronchospasm, with or without urticaria; parenteral intervention indicated; allergy-related edema/angioedema; hypotension
3. Anemia: Hgb <8.0 g/dL and transfusion is indicated.
4. Neutrophil count decrease: <1000 - 500/mm3
5. Lymphocyte count: severe decrease (<500 - 200/mm3) or increase (>20,000/mm3) in blood lymphocytes.
6. Platelet count decrease: <50,000 - 25,000/mm3
7. Nausea: Inadequate oral caloric or fluid intake; tube feeding, total parenteral nutrition (TPN), or hospitalization indicated.
8. Vomiting: ≥ 6 episodes (separated by 5 minutes) in 24 hrs; tube feeding, TPN or hospitalization indicated
9. Diarrhea: Increase of ≥ 7 stools per day over baseline; incontinence; hospitalization indicated; severe increase in ostomy output compared to baseline; limiting self care activities of daily life.
10. Pneumonitis: Sudden worsening of shortness of breath, reduction in pulmonary function tests, new interstitial infiltrates on chest X-ray and fever.

As much as possible data quality is assessed at the data entry point using intelligent on-line data entry via visual basic designed screen forms. Data element constraints, whether independent range and/or format limitations or 'relative' referential integrity limitations, can be enforced by all methods employed for data input. QA reports assess data quality post-data entry. As we note, data quality begins with the design of the data collection forms and procedures and incorporates reasonable checks to minimize transcription and omission errors. Of the more important quality assurance measures are the internal validity checks for reasonableness and consistency.

* Data Monitoring: The DCC identifies missing or unclear data and generates a data query to the consortium administrator contact.
* Data Delinquency Tracking: The Data Coordinating Center will monitor data delinquency on an ongoing basis.

Phase 1b study will require 9 to 15 evaluable subjects. Assuming a 20% drop out rate and 20% screen failure, the target enrollment will be 9-21 subjects. As the primary analysis, the safety data generated from this study will be analyzed to generate an optimum range of dose to be utilized in Phase 2a study. The secondary endpoints will be summarized to help more detailed evaluation in Phase 2a study.

Deviations from the protocol are not allowed. It is the responsibility of each study site to use continuous vigilance to identify and report any protocol deviations. Upon determination that a protocol deviation has occurred, the study staff will a) notify the Principal Investigator, b) notify Project Manager and c) complete the Protocol Deviation form. The Principal Investigator will complete and sign the Protocol Deviation form and submit it to the site Institutional Review Board (IRB), per IRB regulations. Major protocol deviations will be reported to the Data and Safety Monitoring Board. The Investigation New Drug (IND) sponsor will also be informed and will be responsible for notifying the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients. It should be noted, however, that LAM occurs predominantly in women.
* 18 to 65 years of age.
* All patients must have a diagnosis of LAM as defined by one of the following:

Open lung, transbronchial or thoracic needle biopsy consistent with LAM Open or needle abdominal biopsy findings consistent with LAM Computed tomography (CT) of chest or abdomen consistent with LAM in the setting of TSC, renal angiomyolipoma (AML), cystic abdominal lymphangiomas, or history of chylous effusion in the chest or abdomen CT of chest consistent with LAM plus serum vascular endothelial growth factor (VEGF-D) > 800 pg/ml In cases where the diagnosis of LAM is based on biopsy, review of the pathology specimens by pathologists who are experienced with LAM, such as those at the NIH or the Mayo Clinic, will be obtained (if not done so previously).

Exclusion Criteria:

* Current infection.
* Major surgery within the past 2 months
* Advanced hematologic, renal, hepatic, or metabolic diseases
* The use of another investigational drug within 30 days
* The use of mammalian target of rapamycin (mTOR) inhibitors within 30 days
* Previous lung transplantation or active on transplant list.
* Inability to attend scheduled clinic visits
* Inability to give informed consent
* Inability to perform pulmonary function testing
* History of malignancy in the past two years, other than squamous or basal cell skin cancer or mild cervical cancer.
* Nursing mothers
* Current or planned pregnancy.
* Not using adequate contraception (in woman of childbearing potential).
* Significant clinical change in health in the past 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Dose Determination | Saracatinib will be given for 4 weeks, the subject will be followed for a total of 8 weeks.
  One of three escalating daily oral doses of saracatinib; 50, 125 and 175 mg. Saracatinib will be given orally once a day for four weeks. Adverse events will be monitored. The subject will receive only one of the doses as determined by the escalation of the study.

SECONDARY OUTCOMES:
Safety Profile | 8 weeks
  This objective is to generate a safety profile utilizing the data collected along with the adverse events. Subjects will be followed closely during the 4 weeks while taking drug and again for four weeks after stopping the study drug.

OTHER OUTCOMES:
Efficacy exploration | 8 weeks
  explore the efficacy measurements (e.g., pulmonary function test, six minute walk test, and VEGF-D)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Eissa, MD, Study Chair — Baylor College of Medicine; Nicola A Hanania, MD, Principal Investigator — Baylor College of Medicine - Ben Taub Hospital; Khalid Almoosa, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Frank McCormack, MD, Principal Investigator — University of Cincinnati
Locations (3):
- United States (3):
  - University of Cincinnati, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center-Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
The subject is aware of his/her data at the time of the study. They are told if they are/are not using the correct technique for MDI. There is no more data to share with the subject.